CLINICAL TRIAL: NCT07294066
Title: Uniting Trusted Community Messengers to Improve Access to Cervical Cancer Screening in Rural North Carolina Aim 3
Brief Title: Uniting Trusted Community Messengers to Improve Access to Cervical Cancer Screening in Rural North Carolina
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25-1747 Aim3; K23MD020429 (NIH)
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cervix Cancer; Screen HPV-positive
Keywords: Screening; rural; outreach; high risk
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: 100 woman and 12 community partners will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Woman (Experimental): Women living in Lenoir County will receive HPV self-collection with navigation. At the community level, local community-based organizations (CBOs) will serve as human papillomavirus self-collection (HPVSC) kit distribution sites for unscreened or under screened women.
  Interventions: Diagnostic Test: Human papilloma virus screening
- Community partners (No Intervention): Twelve community partners involved in delivering various components of the intervention (e.g., distributing self-collection kits, providing navigation to follow-up care, or providing clinic-based screening for follow-up for HPV positive tests) will complete surveys and interviews to provide feedback about the intervention.

INTERVENTIONS:
Diagnostic Test: Human papilloma virus screening — Human papilloma virus self-collection (HPVSC) kits will be provided to screen HPV.
  Arms: Woman

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of a multi-level, community-engaged intervention to increase access to cervical cancer screening using human papillomavirus (HPV) self-collection (HPVSC) outreach among women living in a high-risk rural county and to improve navigation for follow-up screening.

A one-group intervention evaluation design will be used to pilot test feasibility and acceptability and to assess the proportion of women who return HPVSC kits and test HPV-positive. At the community level, local community-based organizations (CBOs) will serve as HPVSC kit distribution sites. At the individual level, trained community health workers will work with CBOs to support women throughout the HPVSC process, including specimen collection, kit return, result notification, and follow-up clinic-based screening for women who test HPV-positive.

DETAILED DESCRIPTION:
The RE-AIM framework will be applied to selected domains to assess feasibility using predefined parameters. Quantitative surveys will measure acceptability of intervention components among women and community partners, and qualitative interviews will explore their experiences with the intervention.

The RE-AIM framework is a comprehensive tool for evaluating public health and community-based interventions. It focuses on five key dimensions: Reach, which assesses the number, proportion, and representativeness of individuals who participate in a program; Effectiveness, which measures the impact of the intervention on important outcomes, including potential negative effects; Adoption, which examines the number and representativeness of settings or staff that implement the program; Implementation, which evaluates how well the intervention is delivered as intended, including consistency and costs; and Maintenance, which considers the sustainability of both the intervention and its effects over time at individual and organizational levels.

ELIGIBILITY:
Woman participants

Inclusion Criteria:

* Resident of Lenoir County and 12 community.
* have not received a Pap test within the last 3.5 years, or an HPV test in the last 5.5 years
* female ≥ 30 to 64 years of age at time of recruitment

Exclusion Criteria:

* 65 years of age or older had a hysterectomy,
* history of cervical cancer,
* plan to move from Lenoir County during the study period.

Community partners participants

Inclusion Criteria:

* community health workers
* clinic staff
* community-based organization staff.

Exclusion Criteria:

• None

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment and enrollment rate | Up to 6 months
  Proportion of eligible unscreened women recruited, with a target enrollment of 100 participants from Lenoir County.
Retention rate | Up to 6 months
  Ratio of returned HPV self-collection kits to kits distributed, and rate of participant withdrawal or loss to follow-up.
HPV positive screening rate | Up to 6 months
  Rate of HPV-positive screening rate among woman started study will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mansfield, PhD, RN, Principal Investigator — UNC Lineberger Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) generated from this study will be made publicly available. Data will be shared via unrestricted download, with no controlled access. No limitations are anticipated on data access, distribution, or reuse. All shared data will be de-identified to protect participant confidentiality and will be collected and shared in accordance with informed consent, IRB approval, and UNC Research Compliance Program policies.
Time Frame: No later than the time of publication or the end of the funding period, whichever occurs first, and will be preserved for a minimum of 10 years.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials